CLINICAL TRIAL: NCT00533988
Title: Central Venous Catheter-Related Infection: A Prospective Randomized Double-Blind Study
Brief Title: Central Venous Catheter-Related Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Witwatersrand, South Africa (Other)
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: 94/4/4.1;7902114
Record Dates: First submitted 2007-09-21; First posted 2007-09-24 (Estimated); Last update posted 2007-10-01 (Estimated); Status verified 2007-09

CONDITIONS: Critically Ill Patients; Infection
Keywords: Central venous catheters; Antimicrobial impregnated catheters; Duration of catheter use; Catheter-related infection; Insertion site; Parenteral nutrition; Critically ill patients (multidisciplinary)
MeSH Terms: conditions — Infections; Catheter-Related Infections; Hyperphagia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 5592 (No Intervention): Standard triple lumen catheter
- 5593 (Active Comparator): Antimicrobial impregnated catheter (chlorhexidine silver-sulfadiazine)
  Interventions: Device: Antimicrobial impregnated catheter (5593)

INTERVENTIONS:
Device: Antimicrobial impregnated catheter (5593) — Comparison of 14-day placement of a standard triple lumen (ARROW Standard Triple Lumen Catheter, Arrow International Inc., Reading, PA, US) versus an antimicrobial impregnated catheter (Chlorhexidine-silver sulfadiazine)(ARROWgard Triple Lumen Catheter, Arrow International Inc., Reading, PA, US)
  Other Names: ARROW Standard Triple Lumen Catheter; ARROWgard Triple Lumen Catheter
  Arms: 5593

SUMMARY:
Intravascular devices are an integral component of modern-day medical practice. Infection is one of the leading complications of intravascular catheters and is associated with an increased mortality, prolonged hospitalization and increased medical costs. Central venous catheters (CVCs) account for an estimated 90% of all catheter-related bloodstream infections (CRBSI). A host of risk factors for CVC-related infections have been documented. This includes most importantly, duration of catheterization. The duration of use of CVCs remains controversial and the length of time such devices can safely be left in situ has not been fully and objectively addressed in the critically ill patient. As a consequence, scheduled replacement remains widely practiced in many Intensive Care Units(ICUs). Over the past few years, antimicrobial impregnated catheters have been introduced in an attempt to limit catheter-related infection (CRI) and increase the time that CVCs can safely be left in place. Recent meta-analyses concluded that antimicrobial impregnated CVCs appear to be effective in reducing CRI. The topic however, remains extremely controversial with different viewpoints appearing in the literature recently.

This was a prospective randomized double-blind study performed in the multidisciplinary ICU at Johannesburg Hospital over a four year period.The study entailed a comparison of standard triple-lumen versus antimicrobial impregnated CVCs on the rate of CRI. The aim was to determine whether the researchers could safely increase the duration of catheter insertion time from the standard practice of seven days to 14 days, to assess the influence of the antimicrobial impregnated catheter on the incidence of CRI, evaluate risk factors and elucidate the epidemiology of CRI.

DETAILED DESCRIPTION:
Intravascular devices are an integral component of modern-day medical practice. They are used to administer intravenous fluids, medications, blood products and parenteral nutrition. In addition, they serve as a valuable monitor of the hemodynamic status of critically ill patients.

Infection is one of the leading complications of intravascular catheters and is associated with an increased mortality, prolonged hospitalization and increased medical costs. Central venous catheters(CVCs) account for an estimated 90% of all catheter-related bloodstream infections(CRBSI). A host of risk factors for CVC-related infections have been documented. This includes, most importantly, the duration of catheterization. The duration of use of CVCs remains controversial and the length of time such devices can safely be left in situ has not been fully and objectively addressed in the critically ill patient. As a consequence, scheduled replacement remains widely practiced in many Intensive Care Units(ICUs),the mean time in a recent study in mainland Britain, being 6.5 days.Over the past few years, antimicrobial impregnated catheters have been introduced in an attempt to limit catheter-related infection(CRI) and increase the time that CVCs can safely be left in place.Recent meta-analyses concluded that antimicrobial-impregnated CVCs appear to be effective in reducing CRI.The topic remains extremely controversial with differing viewpoints appearing in the literature.

This was a prospective randomized double-blind study performed in the multidisciplinary ICU at Johannesburg Hospital, Johannesburg, South Africa over a four year period. The study included 118 critically ill patients and entailed comparison of a 14-day placement of a standard triple-lumen central venous catheter (ARROW Standard Triple Lumen Catheter, Arrow International Inc., Reading, PA, US) versus an antimicrobial impregnated catheter (chlorhexidine-silver sulfadiazine)(ARROWgard Triple Lumen Catheter, Arrow International Inc.,Reading, PA, US) on the rate of CRI.

The aim was to:

1. Determine whether the duration of catheter insertion time could safely be increased from our standard practice of seven days to fourteen days
2. To assess the influence of the antimicrobial impregnated catheter on the incidence of CRI
3. To evaluate other previously recorded risk factors for CRI, as well as to
4. Elucidate the epidemiology of CRI.

The randomization protocol involved equal numbers of the two types of non-distinguishable catheters being mixed in consignments and then selected in a consecutive fashion for placement in study candidates.

Consent was obtained prior to enrollment in the study. Standard infection control measures were practiced with catheter insertion.

Skin swabs were taken for culture prior to cleansing with a chlorhexidine containing solution and subsequent catheter insertion. Catheters were inspected and dressed daily, and studied for colonization and CRBSI at removal. The origin of each CRBSI was sought by culturing all potential sources (skin, catheter segments, hubs and infusates). A semiquantitative culture of the catheters using the roll-plate technique was performed and DNA-molecular typing employed to assist in microbiological analyses. All relevant clinical data was collected and evaluated.

CRI was defined according to the criteria proposed by the Centers for Disease Control and Prevention in the USA.

The study was approved by the Committee for Research on Human Subjects of the University of the Witwatersrand.

ELIGIBILITY:
Inclusion Criteria:

* critically ill patients likely to require central venous catheter for at least 14 days
* age 18+ years
* white cell count on admission > 4 x 10 to 9/L
* absence of skin burns
* no history of allergy to sulfa containing preparations
* consent obtained
* catheter to be inserted via internal jugular or subclavian veins

Exclusion Criteria:

* age < 18 years
* white blood cell count on admission of less than 4 x 10 to 9/L
* skin burns
* history of allergy to sulfa-containing preparations
* guidewire changes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 1996-01; Study Completion 1999-12 (Actual)

PRIMARY OUTCOMES:
To determine the influence of antimicrobial impregnated catheters on the incidence of catheter-related infection and whether CVCs can safely be left in place for a period of up to 14 days in critically ill patients | 14 days of catheter placement

SECONDARY OUTCOMES:
To elucidate the epidemiology and risks of catheter-related infection in a population of critically ill patients | 14 day catheter placement

CONTACTS AND LOCATIONS:
Overall Officials: Mervyn Mer, MBBChFCP(SA), Principal Investigator — Department of Medicine, Division of Pulmonology and Critical Care, Johannesburg Hospital and University of the Witwatersrand, Johannesburg, South Africa